CLINICAL TRIAL: NCT03599245
Title: A Single Arm, Open Label Multicentre Extension Study To Evaluate The Effectiveness And Safety Of Ocrelizumab In Patients With Multiple Sclerosis Previously Enrolled In A F. Hoffmann-La Roche Sponsored Ocrelizumab Phase IIIb/IV Clinical Trials
Brief Title: This is an Extension Study of the Roche P-trials to Investigate Safety and Effectiveness of Ocrelizumab in Participants With Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN39158; 2017-004886-29 (EudraCT Number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab (Experimental): Participants will receive a single 600-mg infusion of Ocrelizumab every 24 weeks up to Week 72 of this study.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Participants will receive a 600-mg infusion of Ocrelizumab every 24 months for two years.

SUMMARY:
This extension study will evaluate the effectiveness and safety of ocrelizumab in multiple sclerosis (MS) participants who were previously enrolled in a F. Hoffmann-La Roche (Roche) sponsored ocrelizumab phase IIIb/IV trial (i.e. the Parent, P-trial).

DETAILED DESCRIPTION:
This is a single arm, open label, multicenter extension study in participants who completed treatment period with ocrelizumab in the Roche P-trials. Participants will receive treatment with ocrelizumab as single 600 mg infusions every 24 weeks for two years.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Able to comply with the study protocol, in the investigator's judgment
* Completed the treatment period of Roche sponsored ocrelizumab P-trials

Exclusion Criteria:

* Hypersensitivity to ocrelizumab or to any of its excipients.
* Participantss in a severely immunocompromised state until the condition resolves.
* Evidence of any adverse event potentially attributable to ocrelizumab, for which the local label recommends permanent discontinuation.
* Existence of a contra-indication as per SmPC
* Prohibited concomitant medication as specified in protocol
* Participants intending to become pregnant during the study or within 6 months after the last dose of the study drug in the parent study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1055 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Time to onset of CDP sustained for at least 24 weeks and for at least 48 weeks | Up to 2 Years
Percentage of participants who have confirmed disability improvement (CDI), CDP for at least 24 weeks and for at least 48 weeks yearly and over the duration of the treatment | Up to 2 years
Percentage of participants who have improved, stable or worsened disability compared with baseline | Up to 2 years
  Improved, stable or worsened disability is measured by expanded disability status scale (EDSS) (annually/by epoch and over duration of the study) Stable EDSS is defined as EDSS change +/- 0.5. Worsening is > 0.5 increase of EDSS, Improvement is >0.5 decrease of EDSS
Mean change from inclusion in parent study in EDSS score over the course of the treatment | Up to 2 years
Time to 20% increase in timed 25-foot walk test (T25FWT) | Up to 2 years
  Time to 20% increase in timed nine-hole peg test (9HPT) sustained for at least 24 weeks and for at least 48 weeks, and proportion of patients achieving a sustained increase assessed yearly and at the end treatment

SECONDARY OUTCOMES:
Time to first protocol-defined event of disease activity | Up to 2 Years
Time to first relapse | Up to 2 Years
Annualized relapse rate | Up to 2 Years
Percentage of participants relapse free, yearly and over the course of the treatment | Up to 2 Years
Percentage of participants with no evidence of protocol-defined disease activity (NEDA) yearly and over the duration of the treatment | Up to 2 Years
  Disease activity is defined as at least one the following events: protocol-defined relapse; 24 weeks CDP based on increases in EDSS; a T1 Gadolinium (Gd)-enhanced lesion; or a new and/or enlarging T2 hyperintense lesion on magnetic resonance imaging (MRI).
Percentage of participants with no evidence of progression (NEP) | Up to 2 Years
  NEP is defined as no progression sustained for at least 24 weeks on all of the following three components (CDP; 20% increase in timed T25FWT; 20% increase in timed 9HPT yearly and over the course of the treatment
Percentage of participants with no evidence of progression sustained for at least 24 weeks and no active disease (NEPAD) | Up to 2 Years
  NEPAD is defined as no progression on all of the three components of NEP (CDP, T25FWT, 9HPT), no new relapse and no enlarging or new T2 or T1 Gd-enhancing lesion yearly and over the course of the treatment
Change from baseline in cognitive performance as measured by the Symbol digit modalities test (SDMT) | Up to 2 Years
Total number of T1 Gd-enhancing lesions as detected by brain MRI over time | Up to 2 Years
Total number of new and/or enlarging T2 lesion as detected by brain MRI over time | Up to 2 Years
Change in total T1 hypointense lesion volume over time | Up to 2 Years
Total number of fluid-attenuated inversion-recovery (FLAIR) late enhancing lesions as detected by brain MRI over time | Up to 2 Years
Change in brain volume (grey and white matter) as detected by brain MRI over time | Up to 2 Years
Presence and evolution of leptomeningeal follicles as detected by MRI | Up to 2 Years
Time to treatment discontinuation/switch | Up to 2 Years
Participant reported outcomes: Employment status (Work Productivity and Activity Impairment Questionnaire [WPAI]) | Up to 2 Years
Participant reported outcomes: SymptoMScreen Score | Up to 2 Years
Participant reported outcomes: Quality of life (QoL) (Multiple Sclerosis Impact Scale [MSIS]-29) | Up to 2 Years
Percentage of Participants with Adverse Events | Up to 2 Years
Total number of FLAIR late enhancing lesions as detected by brain MRI at the end of the treatment period | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (159):
- Argentina (3):
  - Hospital Churruca Visca, Buenos Aires
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, Ciudad Autonoma Buenos Aires
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
- Belgium (5):
  - AZ Sint Jan, Bruges
  - UZ Antwerpen, Edegem
  - CHU Tivoli, La Louvière
  - CHU de Liège (Sart Tilman), Liège
  - Revalidatie en MS Centrum, Overpelt
- Brazil (3):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Bulgaria (2):
  - Shat Np Sveti Naum, Sofia
  - Multiprofile Hosp. for Active Treatment, Sofia
- Canada (7):
  - University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre Uni Campus, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique NeuroOutaouais, Gatineau, Quebec
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (4):
  - Fakultni nemocnice u sv. Anny, Brno
  - Nemocnice Jihlava, Jihlava
  - VFN Praha Poliklinika Rs Centrum - Budova A, Prague
  - Fakultni nemocnice v Motole, Prague
- Denmark (5):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Odense Universitetshospital, Neurologisk Afdeling N, Odense C
  - Hjerne- og nervesygdomme, Ambulatorium, Skleroseklinikken, Sønderborg
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Mehiläinen Neo Turku, Turku, Finland
- France (17):
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital neurologique Pierre Wertheimer - CHU Lyon, Bron
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH de Gonesse, Gonesse
  - CHU de Grenoble, La Tronche
  - Hopital Roger Salengro Service de Neurologie, Lille
  - CHU de la Timone - Hopital d Adultes, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - Hopital Central - CHU de Nancy, Nancy
  - Hôpital Pasteur, Nice
  - CHU de Nîmes Hopital Caremeau, Nîmes
  - Groupe Hospitalier Pitié- Salpétrière, Paris
  - Hôpital de Poissy, Poissy
  - CHU de Rouen Hopital, Rouen
  - Höpital Hautepierre, Strasbourg
  - HIA de Toulon hôpital militaire, Toulon
- Hungary (2):
  - Budapesti Jahn Ferenc Dél-pesti Kórház és Rendel?intézet, Budapest
  - VALEOMED Diagnosztikai Központ, Esztergom
- St Vincents University Hospital, Dublin, Ireland
- Italy (31):
  - Ospedale SS. Annunziata - Clinica Neurologica - Centro Sclerosi Multipla, Chieti, Abruzzo
  - Ospedale San Salvatore, L’Aquila, Abruzzo
  - IRCCS Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Apulia
  - A. O. U. Federico II, Napoli, Campania
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Ospedale S.Camillo Forlanini, Rome, Lazio
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - ASST PAPA GIOVANNI XXIII Neurologia USS Malattie Autoimmuni Centro Sclerosi Multipla, Bergamo, Lombardy
  - Ospedale S.Antonio Abate, Gallarate, Lombardy
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
  - Ospedale Civile di Montichiari, Montichiari, Lombardy
  - IRCCS Istituto Neurologico C. Mondino?Dip. Neurologia Neuroriabilitazione S.S. Sclerosi Multipla, Pavia, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
  - Ospedale Binaghi, Cagliari, Sardinia
  - AOU Policlinico V. Emanuele - P.O G. Rodolico, Catania, Sicily
  - Fondazione Istituto S. Raffaele - Giglio, Cefalù, Sicily
  - AOU Policlinico Giaccone, Palermo, Sicily
  - AO Ospedali Riuniti Villa Sofia-Cervello, Palermo, Sicily
  - AOU Ospedali Riuniti Umberto I-G.M. Lancisi-G. Salesi, Ancona, The Marches
  - AOU Careggi, Florence, Tuscany
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - AOU Senese - Presidio Ospedaliero Le Scotte, Siena, Tuscany
  - AO di Perugia - Ospedale S. Maria della Misericordia, Perugia, Umbria
  - Azienda Ospedaliera di Padova, Padua, Veneto
  - Policlinico G.B. Rossi, Verona, Veneto
- Ibn Sina Hospital, Kuwait City, Kuwait
- Mexico (3):
  - Hospital General de México, Mexico City, Mexico CITY (federal District)
  - Hospital Angeles de Culiacán, Neurociencias Estudios Clínicos SC, Culiacán, Sinaloa
  - Unidad de investigacion en salud (UIS), Mexico City
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Amsterdam UMC Location VUMC, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Groene Hart Ziekenhuis, Gouda
  - Maasstadziekenhuis, NL -rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
- Norway (3):
  - Haukeland universitetssykehus, Bergen
  - Sykehuset Buskerud HF, Drammen
  - Stavanger Universitetssykehus, Helse Stavanger HF, Stavanger
- Poland (8):
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika, Gdansk
  - Care Clinic, Katowice
  - Malopolskie Centrum Diagnostyczne MEDICAL Sp. z o. o., Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
- Portugal (4):
  - Hospital de Braga, Braga
  - HUC, Coimbra
  - Hospital Beatriz Angelo, Loures
  - Hospital Geral de Santo Antonio, Porto
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Univerzitna nemocnica Bratislava Nemocnica Ruzinov, Bratislava
  - Fakultna nemocnica Trnava, Trnava
- Slovenia (2):
  - University Medical Centre, Ljubljana
  - University Medical Centre Maribor, Maribor
- Spain (17):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Castellon, Castellon, Castellon
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Lerida
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Complejo Hospitalario Universitario de Vigo - Xeral Cies, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Universitario de La Princesa, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario la Fe, Valencia
- Sweden (3):
  - Sahlgrenska Sjukhuset, Gothenburg
  - Centralsjukhuset, Karlstad
  - Centrum för Neurologi, Stockholm
- Turkey (Türkiye) (8):
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Mustafa Kemal Ataturk UTF, Hatay
  - Istanbul University Istanbul School of Medicine, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi, Istanbul
  - Selcuk University Medical Faculty, Konya
  - Ondokuz Mayis University School of Medicine, Samsun
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
- United Kingdom (15):
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Raigmore Hospital, Inverness
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Royal London Hospital, London
  - Royal Free Hospital, London
  - Kings College Hospital, London
  - St George's Hospital, London
  - Charing Cross Hospital, London
  - National Hospital for Neurology and Neurosurgery,, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Salford Royal NHS Foundation Trust, Salford
  - Royal Hallamshire Hospita, Sheffield
  - Morriston Hospital, Swansea
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing